CLINICAL TRIAL: NCT03676244
Title: Immediate Implant Placement With Immediate Provisionalization Into Extraction Sockets With Labial Plate Dehiscence Defects Within the Maxillary Esthetic Zone
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, merna yehia ghoneim, principal investigator, Cairo University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: cairoUimplant program
Record Dates: First submitted 2018-09-16; First posted 2018-09-18 (Actual); Last update posted 2018-09-18 (Actual); Status verified 2018-09

CONDITIONS: Badly Decayed Anterior Maxillary Teeth

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- immediate implant placement in anterior esthetic zone (Experimental): extraction of badly broken anterior maxillary teeth with immediate implant placement
  Interventions: Device: immediate implant in defected anterior maxillary esthetic zone

INTERVENTIONS:
Device: immediate implant in defected anterior maxillary esthetic zone — Patients indicated for immediate implant placement with presence of partial or complete loss (type 2 sockets) of labial bone plate.
  Use of GBR (mix of autogenous bone graft and xenograft in combination to absorbable collagen membrane) and healing abutment at the same time of extraction then place implant palatally engaging the side walls of the socket, leaving a buccal gap.
  construct custom two-piece screw retained healing abutment then remove custom healing abutment and fit and place the collagen membrane for GBR , the membrane should cover the defect 2 mm circumferentially and extend to the level of free gingival margin, Place bone graft material buccal to the implant surface ,replace custom healing abutment.

SUMMARY:
Immediate tooth replacement with implants into extraction sockets has become a common clinical procedure regarding implant survival, osseointegration and esthetics.

Basically, when there is a labial bone plate loss after extraction 2 stage GBR procedure would be carried out to allow adequate amount of bone formation to be reconstructed and receive the dental implant.

The challenge is when there is a partial or complete loss of labial plate of bone resulting from severe trauma or chronic inflammation or vertical fracture affecting the periodontal attachment

DETAILED DESCRIPTION:
Elian etal. classified extraction sockets into 3 types: type 1 sockets have labial plate of bone and soft tissue completely intact, type 2: where the soft tissue is intact while there is a dehiscence bony defect indicating partial or complete loss of labial bone plate, and type 3 where a midfacial recession occurred indicating loss of labial bone plate and soft tissue loss.

The clinical outcomes of type 2 sockets reconstructions: Noelken etal. Published survival of 16 implants immediately placed in sockets with

complete loss of labial bone plate and buccal gaps were filled with autogenous bone without using barrier membrane. IN this study immediate implant is to be placed in type 2 sockets filing the gap with a mix of autogenous bone harvested from tuberosity and xenograft in addition to a resorbable collagen membrane lining the socket and healing abutment .

Immediate implant placement concurrent with provisional restoration has been advocated to improve the esthetic restorative outcome for the patients. The success of this procedure depends on many variables including gingival health and morphology, bone dimensions and primary stability of the implants.

Immediate implant placement is most commonly indicated when tooth extraction is due to trauma,endodontic lesion, root fracture, root resorption, root perforation, unfavorable crown to root ratio(not due to periodontal loss and bony walls

of alveolus are still intact.

Contraindications includes presence of active infection, insufficient bone (<3 mm) beyond the tooth socket apex for initial implant stability and wide and/or long gingival recession.

Immediate implant placement even in the aesthetic zone is a literature supported treatment modality with success comparable to alternative placement protocols.3, 4 Immediate placement reduces the number of surgical interventions, shortens time to final restoration, may offer a fixed provisional restoration alternative to a removable interim prosthesis, and may partially support the peri-implant tissues prior to collapse from the extraction socket remodeling. Certain clinical criteria however need to be met in order to achieve a successful treatment outcome, namely: intact extraction socket walls, facial bone residual at ≥ 1 mm, thick gingival biotype, absence of acute infection, and sufficient residual bone at the palatal and apical tooth socket.

Current knowledge suggests that implant placement should be at least 3 to 4 mm in depth from the midfacial free gingival margin and 2 mm palatally from the facial osseous crest.

ELIGIBILITY:
Inclusion Criteria:

* Patients indicated for immediate implant placement with presence of partial or complete loss (type 2 sockets) of labial bone plate.
* Both sexes.
* No intraoral soft and hard tissue patholog.
* No systemic condition that contraindicate implant placement.

Exclusion Criteria:

* General medical or psychiatric contraindications.
* Pregnancy.
* Patients with local or generalized healing limitations.
* Diabetes.
* Smoking type 3 extraction sockets.
* Bruxism or other Para functional habits.
* Compromised soft tissue conditions.

Ages: 25 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 15 (Estimated)
Dates: Start 2018-09-25 (Estimated); Primary Completion 2019-07 (Estimated); Study Completion 2019-09 (Estimated)

PRIMARY OUTCOMES:
bucco lingual and crestal bone loss | 6 month
  the amount of bone loss will be measured using cone beam computed tomography